CLINICAL TRIAL: NCT06028230
Title: A Parallel-group Treatment, Phase 2, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of SAR444656 in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of SAR444656 Compared With Placebo in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Acronym: ZEN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision. Not related to safety concern.
Sponsor: Sanofi (Industry)
Collaborators: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17841; 2023-504328-25 (Registry Identifier: CTIS); U1111-1285-8790 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR444656 dose 1 (Experimental): Participants will receive SAR444656 dose 1 orally
  Interventions: Drug: SAR444656 (KT-474)
- SAR444656 dose 2 (Experimental): Participants will receive SAR444656 dose 2 orally
  Interventions: Drug: SAR444656 (KT-474)
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR444656 (KT-474) — Oral Tablet
  Arms: SAR444656 dose 1; SAR444656 dose 2
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2, 3-arm study to evaluate the efficacy, safety, PK, and biological effects of SAR444656 compared with placebo in adult participants with moderate to severe HS aged ≥18 to 70 years.

Study details include:

* Screening period: up to 4 weeks (30 days)
* Treatment duration: up to 16 weeks
* Follow-up period: up to 4 weeks
* Total study duration: up to 24 weeks
* Number of visits: 14

ELIGIBILITY:
Inclusion Criteria:

* Participant with a history of signs and symptoms consistent with HS for at least 1 year prior to baseline.
* Participant must have HS lesions present in at least 2 distinct anatomic areas, one of which must be Hurley Stage II or Hurley Stage III.
* Participant must have had an inadequate response after at least one-month of oral antibiotic treatment for HS, as assessed by the Investigator.
* Participant must have a total AN count of ≥5 at the baseline visit.
* Participant must have a draining tunnel count of ≤20 at the baseline visit.
* Participant must be willing and able to complete the diary for the duration of the study as required by the study protocol.
* Contraceptive use by men with a partner of childbearing potential and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Participant with any other active skin disease or condition (eg, bacterial, fungal, or viral infection) that may interfere with assessment of HS.
* Any active or chronic infection requiring systemic treatment (eg, antibiotics, antivirals, antifungals, antihelminthics) within 30 days prior to baseline.
* Known history of or suspected significant suppressed immune response, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Participant with history of solid organ transplant.
* Participant with history of splenectomy.
* Participant with history of any malignancy or lymphoproliferative disease, except if the participant has been free from disease for ≥5 years. Successfully treated non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma, or localized carcinoma in situ of the cervix are allowed.
* Participant with a diagnosis of chronic immune-mediated, inflammatory conditions other than HS
* Participant with family history of sudden death or long QT syndrome.
* Participant with history of congenital or drug-induced long QT syndrome.
* Participant with congestive heart failure (New York Heart Association Class 2 to 4), greater than Class 1 angina pectoris, acute coronary syndrome within prior 6 months, known structural heart disease.
* Participant with history of any major cardiovascular events (eg, myocardial infarction, unstable angina pectoris, coronary revascularization, stroke, or transient ischemic attack) at any time prior to screening.
* Participant with history of ventricular fibrillation, ventricular tachycardia, torsades de pointes, atrial fibrillation, syncope not explained by non-cardiac etiology.
* Participant with uncontrolled hypertension defined as consistent systolic blood pressure ≥150 mmHg or consistent diastolic blood pressure ≥90 mmHg despite antihypertensive medication.
* Participant received prescription topical therapies for the treatment of HS within 14 days prior to the baseline visit.
* Prior or active treatment with any systemic biologic (anti-TNF) therapy, anti-IL17 therapy, anti-IL1/anti-IL1 receptor therapy except for up to 20% of the total study population. Furthermore, this 20% of biologic-experienced participants must fulfilled one or more of the following conditions:

  * Discontinued due to treatment related toxicity and/or
  * Discontinuation is not related to lack or loss of therapeutic response.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in total abscess and inflammatory nodule (AN) count | Week 16
  The AN count is the sum of the abscess count and inflammatory nodule count at any given clinical assessment. It is derived from the lesion counts obtained as part of the HS clinical parameters.

SECONDARY OUTCOMES:
Proportion of participants achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR 50) | Week 16
Proportion of participants achieving AN count ≤2 | Week 16
Absolute change from baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) | Week 16
Proportion of participants with improvement from baseline in Hurley Stage | Week 16
Proportion of participants achieving AN50 (at least 50% reduction in the AN count relative to baseline) | Week 16
Change from baseline in participants reported daily worst pain using HS-Skin Pain-Numerical Rating Scale (HS-Skin Pain-NRS) | Week 16
Proportion of participants achieving improvement defined as at least 30% reduction and at least 1 unit reduction in participant daily worst pain using HS-Skin pain-NRS | Week 16
Change from baseline in the amount of analgesic | Up to Week 16
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs), investigational medicinal product (IMP) discontinuation due to TEAEs | Up to Week 20
Plasma SAR444656 concentration | Up to Week 16

CONTACTS AND LOCATIONS:
Locations (52):
- United States (21):
  - Clear Dermatology & Aesthetics Center- Site Number : 8400006, Scottsdale, Arizona
  - Cosmetic Dermatology of Orange County- Site Number : 8400024, Anaheim, California
  - First OC Dermatology - Fountain Valley- Site Number : 8400007, Fountain Valley, California
  - Paradigm Clinical Research - San Diego - ClinEdge - PPDS- Site Number : 8400021, San Diego, California
  - Clinical Trials Management Services - Thousand Oaks- Site Number : 8400028, Thousand Oaks, California
  - Advanced Dermatology and Cosmetic Care- Site Number : 8400025, Valencia, California
  - Encore Medical Research of Boynton Beach- Site Number : 8400002, Boynton Beach, Florida
  - Moore Clinical Research - Brandon- Site Number : 8400001, Brandon, Florida
  - Encore Medical Research - 6600 Taft St- Site Number : 8400005, Hollywood, Florida
  - Sullivan Dermatology- Site Number : 8400003, Miami, Florida
  - ARA Professionals- Site Number : 8400023, Miami, Florida
  - Encore Medical Research - Weston- Site Number : 8400010, Weston, Florida
  - Dermatology Specialists Research (DS Research) - Indiana- Site Number : 8400012, Clarksville, Indiana
  - Dawes Fretzin Clinical Research- Site Number : 8400011, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center - 110 Francis St- Site Number : 8400013, Boston, Massachusetts
  - Wayne Health - Dearborn- Site Number : 8400004, Dearborn, Michigan
  - Revive Research Institute-1575 W Big Beaver Rd- Site Number : 8400008, Troy, Michigan
  - Vial Health - DermDox Dermatology- Site Number : 8400020, Camp Hill, Pennsylvania
  - Clinical Research Philadelphia,LLC- Site Number : 8400026, Philadelphia, Pennsylvania
  - UPMC Montefiore- Site Number : 8400009, Pittsburgh, Pennsylvania
  - Dermatology Specialists of Spokane- Site Number : 8400015, Spokane, Washington
- Investigational Site Number : 1240004, Québec, Quebec, Canada
- Chile (4):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Independencia
  - Investigational Site Number : 1520001, Las Condes
  - Investigational Site Number : 1520004, Temuco
- Germany (8):
  - Investigational Site Number : 2760002, Heidelberg, Baden-Wurttemberg
  - Investigational Site Number : 2760008, Munich, Bavaria
  - Investigational Site Number : 2760006, Würzburg, Bavaria
  - Investigational Site Number : 2760007, Frankfurt am Main, Hesse
  - Investigational Site Number : 2760001, Bochum, North Rhine-Westphalia
  - Investigational Site Number : 2760004, Remscheid, North Rhine-Westphalia
  - Investigational Site Number : 2760009, Dessau, Saxony-Anhalt
  - Investigational Site Number : 2760005, Berlin
- Greece (3):
  - Investigational Site Number : 3000003, Athens, Attica
  - Investigational Site Number : 3000001, Pavlos Melas, Thessaloniki
  - Investigational Site Number : 3000002, Thessaloniki
- Poland (6):
  - Investigational Site Number : 6160006, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160002, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160005, Lodz, Lódzkie
  - Investigational Site Number : 6160003, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160007, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160004, Ossy, Silesian Voivodeship
- South Korea (4):
  - Investigational Site Number : 4100002, Cheonan-si, Chungcheongnam-do
  - Investigational Site Number : 4100001, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100003, Seongbuk-Gu, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 7240004, Cadiz, Cádiz
  - Investigational Site Number : 7240005, Manises, Valencia
  - Investigational Site Number : 7240003, Alicante
  - Investigational Site Number : 7240001, Granada
  - Investigational Site Number : 7240002, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17841 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25558&tenant=MT_SNY_9011